CLINICAL TRIAL: NCT03535727
Title: A Phase I/II Study of Gemcitabine, Nab-paclitaxel, Capecitabine, Cisplatin, and Irinotecan (GAX-CI) in Combination in Metastatic Pancreatic Cancer
Brief Title: A Study of Gemcitabine, Nab-paclitaxel, Capecitabine, Cisplatin, and Irinotecan in Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J1847; IRB00167664 (Other: Johns Hopkins Medical Institution)
Record Dates: First submitted 2018-05-11; First posted 2018-05-24 (Actual); Results first posted 2024-01-08 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Adenocarcinoma; Pancreatic Neoplasms; Neoplasm, Glandular; Neoplasms; Neoplasms Pancreatic; Digestive System Neoplasm; Endocrine Gland Neoplasms; Digestive System Disease; Pancreatic Diseases; Endocrine System Diseases
MeSH Terms: conditions — Adenocarcinoma; Pancreatic Neoplasms; Neoplasms, Glandular and Epithelial; Neoplasms; Digestive System Neoplasms; Endocrine Gland Neoplasms; Digestive System Diseases; Pancreatic Diseases; Endocrine System Diseases | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine; Capecitabine; Cisplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Phase 1, Cohort 1, Dose level 1 (Experimental): Gemcitabine: 500 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Nab-paclitaxel: 40 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Capecitabine: 500 mg BID, PO twice daily (BID); Days 1-7, 15-21 of a 28 day cycle
  Cisplatin: 20 mg/m^2, IV over 60 minutes; Days 1 and 15 of a 28 day cycle
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Capecitabine; Drug: Cisplatin; Drug: Irinotecan
- Phase 1, Cohort 1, Dose level 2 (Experimental): Gemcitabine 500 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Nab-paclitaxel 60 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Capecitabine: 500 mg BID: PO twice daily (BID); Days 1-7, 15-21 of a 28 day cycle
  Cisplatin: 20 mg/m^2, IV over 60 minutes; Days 1 and 15 of a 28 day cycle
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Capecitabine; Drug: Cisplatin; Drug: Irinotecan
- Phase 1, Cohort 1, Dose level 3 (Experimental): Gemcitabine: 500 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Nab-paclitaxel: 80 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Capecitabine: 500 mg BID, PO twice daily (BID); Days 1-7, 15-21 of a 28 day cycle
  Cisplatin 20 mg/m^2, IV over 60 minutes; Days 1 and 15 of a 28 day cycle
  Irinotecan:20 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Capecitabine; Drug: Cisplatin; Drug: Irinotecan
- Phase 1, Cohort 1, Dose level 4 (Experimental): Gemcitabine:500 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Nab-paclitaxel:100 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Capecitabine:500 PO twice daily (BID); Days 1-7, 15-21 of a 28 day cycle
  Cisplatin:20 mg/m^2, IV over 60 minutes; Days 1 and 15 of a 28 day cycle
  Irinotecan:20 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Capecitabine; Drug: Cisplatin; Drug: Irinotecan
- Phase 1, Cohort 1, Dose level 5 (Experimental): Gemcitabine:500 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Nab-paclitaxel:125 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Capecitabine: 500 mg BID, PO twice daily (BID); Days 1-7, 15-21 of a 28 day cycle
  Cisplatin:20 mg/m^2, IV over 60 minutes; Days 1 and 15 of a 28 day cycle
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Capecitabine; Drug: Cisplatin; Drug: Irinotecan
- Phase 1, Cohort 2, Dose level 1 (Experimental): Gemcitabine: 500 mg/m^2, IV over 30 minutes; Days 4 and 11 of a 21 day cycle
  Nab-paclitaxel:40 mg/m^2, IV over 30 minutes; Days 4 and 11 of a 21 day cycle
  Capecitabine:500 mg BID, PO twice daily (BID); Days 1-14 of a 21 day cycle
  Cisplatin:20 mg/m^2, IV over 60 minutes; Days 4 and 11 of a 21 day cycle
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 4 and 11 of a 21 day cycle
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Capecitabine; Drug: Cisplatin; Drug: Irinotecan
- Phase 1, Cohort 2, Dose level 2 (Experimental): Gemcitabine: 500 mg/m^2, IV over 30 minutes; Days 4 and 11 of a 21 day cycle
  Nab-paclitaxel:60 mg/m^2, IV over 30 minutes; Days 4 and 11 of a 21 day cycle
  Capecitabine:500mg BID, PO twice daily (BID); Days 1-14 of a 21 day cycle
  Cisplatin:20 mg/m^2, IV over 60 minutes; Days 4 and 11 of a 21 day cycle
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 4 and 11 of a 21 day cycle
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Capecitabine; Drug: Cisplatin; Drug: Irinotecan
- Phase 1, Cohort 2, Dose level 3 (Experimental): Gemcitabine: 500 mg/m^2, IV over 30 minutes; Days 4 and 11 of a 21 day cycle
  Nab-paclitaxel:80 mg/m^2, IV over 30 minutes; Days 4 and 11 of a 21 day cycle
  Capecitabine:500mg BID, PO twice daily (BID); Days 1-14 of a 21 day cycle
  Cisplatin:20 mg/m^2, IV over 60 minutes; Days 4 and 11 of a 21 day cycle
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 4 and 11 of a 21 day cycle
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Capecitabine; Drug: Cisplatin; Drug: Irinotecan
- Phase 2 Dose Expansion (Cohort 1, DL5) (Experimental): Gemcitabine:500 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Nab-paclitaxel:125 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Capecitabine: 500 mg BID, PO twice daily (BID); Days 1-7, 15-21 of a 28 day cycle
  Cisplatin:20 mg/m^2, IV over 60 minutes; Days 1 and 15 of a 28 day cycle
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Capecitabine; Drug: Cisplatin; Drug: Irinotecan

INTERVENTIONS:
Drug: Nab-paclitaxel — IV over 30 minutes; Days 1 and 15
  Other Names: Abraxane
  Arms: Phase 1, Cohort 1, Dose level 1; Phase 1, Cohort 1, Dose level 2; Phase 1, Cohort 1, Dose level 3; Phase 1, Cohort 1, Dose level 4; Phase 1, Cohort 1, Dose level 5; Phase 2 Dose Expansion (Cohort 1, DL5)
Drug: Gemcitabine — IV over 30 minutes; Days 1 and 15
  Other Names: Gemzar
  Arms: Phase 1, Cohort 1, Dose level 1; Phase 1, Cohort 1, Dose level 2; Phase 1, Cohort 1, Dose level 3; Phase 1, Cohort 1, Dose level 4; Phase 1, Cohort 1, Dose level 5; Phase 2 Dose Expansion (Cohort 1, DL5)
Drug: Capecitabine — PO twice daily (BID); Days 1-7, 15-21
  Other Names: Xeloda
  Arms: Phase 1, Cohort 1, Dose level 1; Phase 1, Cohort 1, Dose level 2; Phase 1, Cohort 1, Dose level 3; Phase 1, Cohort 1, Dose level 4; Phase 1, Cohort 1, Dose level 5; Phase 2 Dose Expansion (Cohort 1, DL5)
Drug: Cisplatin — IV over 60 minutes; Days 1 and 15
  Other Names: Platinol
  Arms: Phase 1, Cohort 1, Dose level 1; Phase 1, Cohort 1, Dose level 2; Phase 1, Cohort 1, Dose level 3; Phase 1, Cohort 1, Dose level 4; Phase 1, Cohort 1, Dose level 5; Phase 2 Dose Expansion (Cohort 1, DL5)
Drug: Irinotecan — IV over 30 minutes; Days 1 and 15
  Other Names: Camptosar
  Arms: Phase 1, Cohort 1, Dose level 1; Phase 1, Cohort 1, Dose level 2; Phase 1, Cohort 1, Dose level 3; Phase 1, Cohort 1, Dose level 4; Phase 1, Cohort 1, Dose level 5; Phase 2 Dose Expansion (Cohort 1, DL5)
Drug: Nab-paclitaxel — IV over 30 minutes; Days 4 and 11
  Other Names: Abraxane
  Arms: Phase 1, Cohort 2, Dose level 1; Phase 1, Cohort 2, Dose level 2; Phase 1, Cohort 2, Dose level 3
Drug: Gemcitabine — IV over 30 minutes; Days 4 and 11
  Other Names: Gemzar
  Arms: Phase 1, Cohort 2, Dose level 1; Phase 1, Cohort 2, Dose level 2; Phase 1, Cohort 2, Dose level 3
Drug: Capecitabine — PO BID; Days 1- 14
  Other Names: Xeloda
  Arms: Phase 1, Cohort 2, Dose level 1; Phase 1, Cohort 2, Dose level 2; Phase 1, Cohort 2, Dose level 3
Drug: Cisplatin — IV over 60 minutes; Days 4 and 11
  Other Names: Platinol
  Arms: Phase 1, Cohort 2, Dose level 1; Phase 1, Cohort 2, Dose level 2; Phase 1, Cohort 2, Dose level 3
Drug: Irinotecan — IV over 30 minutes; Days 4 and 11
  Other Names: Camptosar
  Arms: Phase 1, Cohort 2, Dose level 1; Phase 1, Cohort 2, Dose level 2; Phase 1, Cohort 2, Dose level 3

SUMMARY:
The purpose of this study is to evaluate the clinical activity of gemcitabine, nab-paclitaxel, capecitabine, cisplatin, and irinotecan (GAX-CI) in patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This was a two-part, single-institution, open-label, dose-escalation, phase 1/2 study to evaluate the clinical activity of gemcitabine, nab-paclitaxel, capecitabine, cisplatin, and irinotecan in patients with metastatic pancreatic cancer.

Part 1 of the study was a Phase 1 3 + 3 dose escalation study designed to evaluate the maximally tolerated dose (MTD) and safety of increasing doses of nab-paclitaxel in combination with gemcitabine, capecitabine, cisplatin, and irinotecan. There were two cohorts of dose escalations. The two cohorts differed based on the treatment cycle length (28 days for Cohort 1 and 21 days for Cohort 2). Dose escalation started with Cohort 1. Enrollment for Cohort 2 dose level 1 began once dose level 2 of Cohort 1 was shown to be safe and did not exceed MTD.

Part 2 was a Phase 2 expansion cohort study for the evaluation of efficacy once the MTD had been determined.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed untreated metastatic pancreatic adenocarcinoma.
* Patients with the presence of at least one measurable lesion.
* Male or non-pregnant and non-lactating female of age >18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests.
* Must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who will be considered for surgery are ineligible.
* Patient who have had any prior chemotherapy within 5 years of enrollment.
* Patient who have had radiotherapy for pancreatic cancer.
* Age ≥ 76 years
* Patient who is receiving or have received any other investigational agents within 28 days prior to Day 1 of treatment in this study.
* Patient who has undergone major surgery, other than diagnostic surgery within 28 days prior to Day 1 of treatment in this study.
* Patient who has known brain metastases.
* Patient with history of hypersensitivity or allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine, nab-paclitaxel, capecitabine, cisplatin, or irinotecan.
* Patient with uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patient who has serious medical risk factors involving any of the major organ systems.
* Patient who has known history of infection with HIV, hepatitis B, or hepatitis C.
* Pregnant or breast feeding.
* Patient is unwilling or unable to comply with study procedures
* Patient with clinically significant wound.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dung Le, MD, Principal Investigator — Johns Hopkins Medical Institution
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 2 MTD Dose Expansion: Gemcitabine:500 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Nab-paclitaxel:125 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Capecitabine: 500 mg BID, PO twice daily (BID); Days 1-7, 15-21 of a 28 day cycle
  Cisplatin:20 mg/m^2, IV over 60 minutes; Days 1 and 15 of a 28 day cycle
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
Period: Overall Study
Arm/Group | Phase 1, Cohort 1, Dose Level 1 | Phase 1, Cohort 1, Dose Level 2 | Phase 1, Cohort 1, Dose Level 3 | Phase 1, Cohort 1, Dose Level 4 | Phase 1, Cohort 1, Dose Level 5 | Phase 1, Cohort 2, Dose Level 1 | Phase 1, Cohort 2, Dose Level 2 | Phase 1, Cohort 2, Dose Level 3 | Phase 2 MTD Dose Expansion
Started | 3 | 6 | 6 | 6 | 6 | 3 | 3 | 7 | 8
Completed | 3 | 6 | 6 | 6 | 6 | 3 | 3 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1, Cohort 1, Dose Level 2: Gemcitabine: 500 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Nab-paclitaxel: 60 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Capecitabine: 500 mg BID, PO twice daily (BID); Days 1-7, 15-21 of a 28 day cycle
  Cisplatin: 20 mg/m^2, IV over 60 minutes; Days 1 and 15 of a 28 day cycle
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
- Phase 1, Cohort 1, Dose Level 3: Gemcitabine: 500 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Nab-paclitaxel: 80 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Capecitabine: 500 mg BID, PO twice daily (BID); Days 1-7, 15-21 of a 28 day cycle
  Cisplatin: 20 mg/m^2, IV over 60 minutes; Days 1 and 15 of a 28 day cycle
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
- Phase 1, Cohort 1, Dose Level 4: Gemcitabine: 500 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Nab-paclitaxel: 100 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Capecitabine: 500 mg BID, PO twice daily (BID); Days 1-7, 15-21 of a 28 day cycle
  Cisplatin: 20 mg/m^2, IV over 60 minutes; Days 1 and 15 of a 28 day cycle
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
- Phase 1, Cohort 1, Dose Level 5; Phase 2, MTD Dose Expansion: Gemcitabine: 500 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Nab-paclitaxel: 125 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Capecitabine: 500 mg BID, PO twice daily (BID); Days 1-7, 15-21 of a 28 day cycle
  Cisplatin: 20 mg/m^2, IV over 60 minutes; Days 1 and 15 of a 28 day cycle
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
- Phase 1, Cohort 2, Dose Level 2: Gemcitabine: 500 mg/m^2, IV over 30 minutes; Days 4 and 11 of a 21 day cycle
  Nab-paclitaxel:60 mg/m^2, IV over 30 minutes; Days 4 and 11 of a 21 day cycle
  Capecitabine:500 mg BID, PO twice daily (BID); Days 1-14 of a 21 day cycle
  Cisplatin:20 mg/m^2, IV over 60 minutes; Days 4 and 11 of a 21 day cycle
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 4 and 11 of a 21 day cycle
- Phase 1, Cohort 2, Dose Level 3: Gemcitabine: 500 mg/m^2, IV over 30 minutes; Days 4 and 11 of a 21 day cycle
  Nab-paclitaxel:80 mg/m^2, IV over 30 minutes; Days 4 and 11 of a 21 day cycle
  Capecitabine:500 mg BID, PO twice daily (BID); Days 1-14 of a 21 day cycle
  Cisplatin:20 mg/m^2, IV over 60 minutes; Days 4 and 11 of a 21 day cycle
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 4 and 11 of a 21 day cycle
- Total: Total of all reporting groups
Arm/Group | Phase 1, Cohort 1, Dose Level 1 | Phase 1, Cohort 1, Dose Level 2 | Phase 1, Cohort 1, Dose Level 3 | Phase 1, Cohort 1, Dose Level 4 | Phase 1, Cohort 1, Dose Level 5 | Phase 1, Cohort 2, Dose Level 1 | Phase 1, Cohort 2, Dose Level 2 | Phase 1, Cohort 2, Dose Level 3 | Phase 2, MTD Dose Expansion | Total
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 3 | 3 | 7 | 8 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 2 | 5 | 3 | 2 | 1 | 7 | 4 | 27
  >=65 years | 2 | 4 | 4 | 1 | 3 | 1 | 2 | 0 | 4 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 3 | 3 | 2 | 2 | 0 | 4 | 5 | 25
  Male | 1 | 2 | 3 | 3 | 4 | 1 | 3 | 3 | 3 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 6 | 6 | 6 | 6 | 3 | 3 | 7 | 8 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 6
  White | 3 | 6 | 5 | 4 | 6 | 2 | 2 | 6 | 6 | 40
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 6 | 6 | 6 | 6 | 3 | 3 | 7 | 8 | 48
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — The ECOG scale measures performance status , which scores ranging from 0-5: 0=fully active , performs without restrictions, 1=can ambulate,but restricted in physical strenuous activity,2=ambulatory and capable of self care , but unable to work , active for >50%of waking hours,3=limited self care, confined to bed or chair for >50%of waking hours,4=completely disabled, totally confined tp bed/chair,5= deceased
  Participants
    ECOG 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 6
    ECOG 1 | 3 | 5 | 6 | 5 | 6 | 2 | 3 | 5 | 7 | 42

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Gemcitabine.
Description: Dose escalation (phase I portion of the trial only) to determine the MTD in mg/m^2. Participants received Gemcitabine: 500 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle (Cohort 1) or Days 4 and 11 of a 21 day cycle (Cohort 2)
Time Frame: 28 days
Population: Cohort 1 cycle schedule was selected for the MTD (Days 1 and 15 of a 28 day cycle)
Measure: Number; unit: mg/m^2
Groups:
- Phase I: Gemcitabine:500 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle (Cohort 1) or Days 4 and 11 of a 21 day cycle (Cohort 2)
  Nab-paclitaxel:20, 40, 60, 80, 100,125 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle (Cohort 1) or Days 4 and 11 of a 21 day cycle (Cohort 2)
  Capecitabine: 500 mg BID, PO twice daily (BID); Days 1-7, 15-21 of a 28 day cycle (Cohort 1) or Days 1-14 of a 21 day cycle (Cohort 2)
  Cisplatin:20 mg/m^2, IV over 60 minutes; Days 1 and 15 of a 28 day cycle (Cohort 1) or Days 4 and 11 of a 21 day cycle (Cohort 2)
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle (Cohort 1) or Days 4 and 11 of a 21 day cycle (Cohort 2)
Arm/Group | Phase I
Number analyzed (Participants) | 40
mg/m^2 | 500

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Nab-paclitaxel.
Description: Dose escalation (phase I portion of the trial only) to determine the MTD in mg/m^2. Participants received Nab-paclitaxel: 20, 40, 60, 80, 100,125 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle (Cohort 1) or Days 4 and 11 of a 21 day cycle (Cohort 2)
Time Frame: 28 days
Population: Cohort 1 cycle schedule was selected for the MTD (Days 1 and 15 of a 28 day cycle)
Measure: Number; unit: mg/m^2
Groups:
- Phase 1: Gemcitabine:500 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle (Cohort 1) or Days 4 and 11 of a 21 day cycle (Cohort 2)
  Nab-paclitaxel:20, 40, 60, 80, 100,125 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle (Cohort 1) or Days 4 and 11 of a 21 day cycle (Cohort 2)
  Capecitabine: 500 mg BID, PO twice daily (BID); Days 1-7, 15-21 of a 28 day cycle (Cohort 1) or Days 1-14 of a 21 day cycle (Cohort 2)
  Cisplatin:20 mg/m^2, IV over 60 minutes; Days 1 and 15 of a 28 day cycle cycle (Cohort 1) or Days 4 and 11 of a 21 day cycle (Cohort 2)
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle (Cohort 1) or Days 4 and 11 of a 21 day cycle (Cohort 2)
Arm/Group | Phase 1
Number analyzed (Participants) | 40
mg/m^2 | 125

3. Primary Outcome: Maximum Tolerated Dose (MTD) of Capecitabine.
Description: Dose escalation (phase I portion of the trial only) to determine the MTD in mg for twice daily (BID) use. Participants received Capecitabine: 500 mg BID, PO twice daily (BID); Days 1-7, 15-21 of a 28 day cycle (Cohort 1) or Days 1-14 of a 21 day cycle (Cohort 2)
Time Frame: 28 days
Population: Cohort 1 cycle schedule was selected for the MTD (Days 1-7 and 15-21 of a 28 day cycle)
Measure: Number; unit: mg BID
Arm/Group | Phase I
Number analyzed (Participants) | 40
mg BID | 500

4. Primary Outcome: Maximum Tolerated Dose (MTD) of Cisplatin.
Description: Dose escalation (phase I portion of the trial only) to determine the MTD in mg/m^2. Participants received Cisplatin:20 mg/m^2, IV over 60 minutes; Days 1 and 15 of a 28 day cycle (Cohort 1) or Days 4 and 11 of a 21 day cycle (Cohort 2)
Time Frame: 28 days
Population: Cohort 1 cycle schedule was selected for the MTD (Days 1 and 15 of a 28 day cycle)
Measure: Number; unit: mg/m^2
Groups:
- Phase 1: Gemcitabine:500 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle (Cohort 1) or Days 4 and 11 of a 21 day cycle (Cohort 2)
  Nab-paclitaxel:20, 40, 60, 80, 100,125 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle (Cohort 1) or Days 4 and 11 of a 21 day cycle (Cohort 2)
  Capecitabine: 500 mg BID, PO twice daily (BID); Days 1-7, 15-21 of a 28 day cycle (Cohort 1) or Days 1-14 of a 21 day cycle (Cohort 2)
  Cisplatin:20 mg/m^2, IV over 60 minutes; Days 1 and 15 of a 28 day cycle (Cohort 1) or Days 4 and 11 of a 21 day cycle (Cohort 2)
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle (Cohort 1) or Days 4 and 11 of a 21 day cycle (Cohort 2)
Arm/Group | Phase 1
Number analyzed (Participants) | 40
mg/m^2 | 20

5. Primary Outcome: Maximum Tolerated Dose (MTD) of Irinotecan.
Description: Dose escalation (phase I portion of the trial only) to determine the MTD in mg/m^2. Participants received Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle (Cohort 1) or Days 4 and 11 of a 21 day cycle (Cohort 2)
Time Frame: 28 days
Population: Cohort 1 cycle schedule was selected for the MTD (Days 1 and 15 of a 28 day cycle)
Measure: Number; unit: mg/m^2
Arm/Group | Phase 1
Number analyzed (Participants) | 40
mg/m^2 | 20

6. Primary Outcome: Progression-free Survival (PFS) Using RECIST 1.1 Criteria
Description: PFS is defined as the number of months from the date of first dose to disease progression (progressive disease [PD] or relapse from complete response [CR] as assessed using RECIST 1.1 criteria) or death due to any cause. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on the Kaplan-Meier curve.
Time Frame: 27 months
Population: Per the clinical trial design, PFS analyses included all subjects who received the MTD (Cohort 1, Dose Level 5). Since the enrollment criteria and dose are the same, combining those who are treated at MTD at both phases increase the power and enable to estimate the treatment effect with increased precision. This included the 6 subjects enrolled in the Phase 1 portion of the trial and the 8 subjects enrolled in the Phase 2 portion of the trial for a total of 14 subjects.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase 1 MTD/ Phase 2: Gemcitabine:500 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Nab-paclitaxel:125 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Capecitabine: 500 mg BID, PO twice daily (BID); Days 1-7, 15-21 of a 28 day cycle
  Cisplatin:20 mg/m^2, IV over 60 minutes; Days 1 and 15 of a 28 day cycle
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
Arm/Group | Phase 1 MTD/ Phase 2
Number analyzed (Participants) | 14
months | 5.92 [5.52 to NA] — Insufficient number of patients with events.

7. Secondary Outcome: Safety of the Combination of Gemcitabine, Nab-paclitaxel, Capecitabine, Cisplatin, and Irinotecan (GAX-CI) in Patients With Untreated Metastatic PDA.
Description: Number of patients who received the MTD (Cohort 1, Dose Level 5) that experienced a limiting toxicity. Limiting toxicity was defined as a grade 3 or above treatment-related toxicity, with the following exceptions: 1. Grade 3 anemia that resolves to < grade 2 within 7 days; 2. Grade 3 thrombocytopenia without clinically significant bleeding that resolves to < grade 2 within 7 days; 3. Grade 3 or 4 neutropenia that resolves to <grade 2 within 7 days; 4. Grade 3 or 4 leucopenia/lymphopenia; 5. Grade 3 nausea, vomiting, or diarrhea that resolves to <grade 2 within 72 hours; 6. Grade 3 or 4 asymptomatic laboratory values that resolve to < grade 2 within 7 days; 7. Grade 3 dermatologic AEs that are considered mild in severity but only considered grade 3 because of >30% body surface involvement; 8. Grade 3 fatigue lasting less than 72 hours. This study used the descriptions and grading scales found in the revised NCI CTCAE fV 5.0 for adverse event reporting.
Time Frame: 27 months
Population: Per the clinical trial design, safety analyses included all subjects who received the MTD (Cohort 1, Dose Level 5). Since the enrollment criteria and dose are the same, combining those who are treated at MTD at both phases enable to estimate the toxicity rate with increased precision. This included the 6 subjects enrolled in the Phase 1 portion of the trial and the 8 subjects enrolled in the Phase 2 portion of the trial for a total of 14 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 MTD/ Phase 2
Number analyzed (Participants) | 14
Participants | 3

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was assessed for up to 51 months for patients in both Phase 1 and Phase 2 portions of the trial. Serious and Other (Not Including Serious) Adverse Events were assessed up to 45 months for patients in both Phase 1 and 2 portions of the trial.
Description: This study used the descriptions and grading scales found in the revised National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 for adverse event reporting. During the survival follow-up portion of the trial, patients were evaluated for all-cause mortality past the time frame for treatment and the assessment of adverse events.
Groups:
- Phase 1, Cohort 1, Dose Level 1: Gemcitabine: 500 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Nab-paclitaxel: 40 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Capecitabine: 500 mg BID, PO twice daily (BID); Days 1-7, 15-21 of a 28 day cycle
  Cisplatin: 20 mg/^2, IV over 60 minutes; Days 1 and 15 of a 28 day cycle
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
- Phase 2 MTD Dose Expansion: Gemcitabine: 500 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Nab-paclitaxel: 125 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
  Capecitabine: 500 mg BID, PO twice daily (BID); Days 1-7, 15-21 of a 28 day cycle
  Cisplatin: 20 mg/m^2, IV over 60 minutes; Days 1 and 15 of a 28 day cycle
  Irinotecan: 20 mg/m^2, IV over 30 minutes; Days 1 and 15 of a 28 day cycle
Arm/Group | Phase 1, Cohort 1, Dose Level 1 | Phase 1, Cohort 1, Dose Level 2 | Phase 1, Cohort 1, Dose Level 3 | Phase 1, Cohort 1, Dose Level 4 | Phase 1, Cohort 1, Dose Level 5 | Phase 1, Cohort 2, Dose Level 1 | Phase 1, Cohort 2, Dose Level 2 | Phase 1, Cohort 2, Dose Level 3 | Phase 2 MTD Dose Expansion
All-Cause Mortality (participants affected / at risk) | 3/3 | 6/6 | 5/6 | 6/6 | 6/6 | 3/3 | 3/3 | 7/7 | 7/8
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/6 | 5/6 | 2/6 | 4/6 | 1/3 | 2/3 | 2/7 | 4/8
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 6/6 | 6/6 | 6/6 | 3/3 | 3/3 | 7/7 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Cohort 1, Dose Level 1 (N=3) | Phase 1, Cohort 1, Dose Level 2 (N=6) | Phase 1, Cohort 1, Dose Level 3 (N=6) | Phase 1, Cohort 1, Dose Level 4 (N=6) | Phase 1, Cohort 1, Dose Level 5 (N=6) | Phase 1, Cohort 2, Dose Level 1 (N=3) | Phase 1, Cohort 2, Dose Level 2 (N=3) | Phase 1, Cohort 2, Dose Level 3 (N=7) | Phase 2 MTD Dose Expansion (N=8)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disease progression-Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudocyst infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Cohort 1, Dose Level 1 (N=3) | Phase 1, Cohort 1, Dose Level 2 (N=6) | Phase 1, Cohort 1, Dose Level 3 (N=6) | Phase 1, Cohort 1, Dose Level 4 (N=6) | Phase 1, Cohort 1, Dose Level 5 (N=6) | Phase 1, Cohort 2, Dose Level 1 (N=3) | Phase 1, Cohort 2, Dose Level 2 (N=3) | Phase 1, Cohort 2, Dose Level 3 (N=7) | Phase 2 MTD Dose Expansion (N=8)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (13) | 3 (9) | 1 (2) | 2 (11) | 2 (11) | 2 (24) | 6 (21) | 1 (1)
Swollen gland (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 2 (3) | 3 (3) | 3 (4) | 3 (5) | 3 (15) | 4 (14) | 2 (2)
Feeling of water/air in right ear (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyromegaly (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital edema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision decreased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Double vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival chalsis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient eye yellowing (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (4) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (4) | 2 (2) | 5 (7) | 2 (2) | 3 (6) | 4 (7) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 3 (4) | 3 (6) | 2 (3) | 2 (2) | 2 (3) | 3 (3) | 5 (5)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (5) | 4 (4) | 1 (1) | 2 (2) | 2 (3) | 2 (2)
Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White coating on tongue (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Discolored tongue (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue swollen (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Black stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Early satiety (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stool discoloration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dumping after meals (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stools light and floating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased saliva (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 2 (2)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (3) | 3 (4) | 3 (3) | 1 (1) | 4 (6) | 3 (5) | 2 (2) | 2 (3) | 2 (2)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (3) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Fever (General disorders) | 0 (0) | 1 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatosplenomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver Cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (4) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 3 (3) | 1 (1) | 2 (7) | 1 (2) | 2 (2)
Fracture spinal (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 3 (3) | 1 (2) | 1 (5) | 1 (5) | 0 (0)
International Normalized Ratio increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cocaine metabolite (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (10) | 1 (1) | 3 (6) | 1 (1) | 2 (19) | 3 (4) | 2 (5)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 1 (6) | 1 (1) | 1 (1) | 3 (10) | 2 (5) | 3 (11) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 2 (7) | 3 (7) | 1 (2) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight gain (Investigations) | 1 (2) | 3 (8) | 2 (5) | 2 (2) | 2 (4) | 3 (9) | 1 (1) | 2 (5) | 2 (3)
Weight loss (Investigations) | 0 (0) | 2 (3) | 3 (5) | 3 (5) | 4 (6) | 2 (2) | 3 (11) | 3 (6) | 2 (4)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 2 (3) | 2 (7) | 1 (1) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperkalemia (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (6) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 2 (5) | 0 (0) | 2 (2) | 0 (0) | 1 (4) | 2 (3) | 3 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 4 (13) | 4 (5) | 1 (2) | 4 (7) | 1 (1) | 3 (11) | 4 (5) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 1 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 2 (3) | 2 (4) | 1 (1) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Pseudo gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaw pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremities (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (4) | 2 (3) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Neoplasms Benign, Malignant and Unspecified (Incl Cysts and Polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Concentration impairment (Nervous system disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 3 (4) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aura (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sensitivity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jitteriness (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye twitch (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (4) | 3 (4) | 3 (5) | 3 (3) | 3 (3) | 2 (4) | 4 (6) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Confusion (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Insomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal cysts (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal dysfunction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 2 (3) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 3 (4) | 1 (1) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 2 (3) | 2 (2) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus drainage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 2 (2) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 4 (5) | 5 (5) | 5 (6) | 1 (1) | 1 (1) | 6 (6) | 4 (5)
Dry skin (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (4) | 4 (8) | 1 (2)
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipoma and other skin nodules (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arterial thromboembolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (3) | 0 (0) | 1 (3) | 2 (2) | 4 (5) | 2 (7) | 1 (9) | 2 (7) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 3 (4) | 2 (4) | 2 (4) | 2 (3) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 2 (3) | 2 (2) | 1 (1) | 2 (2)
Fungal foot Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cold sore (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sternal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasions and injuries (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash acne form (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Redness and skin sensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Venous stasis dermatitis of lower extremities (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drop foot (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT03535727/Prot_SAP_000.pdf